CLINICAL TRIAL: NCT07351721
Title: Borrelia Arthritis - a Hidden Cause of Arthritis in Danish Patients? Sub-study 1:Incidence&Outcomes Sub-study 2:Characterisation
Brief Title: Borrelia Arthritis - a Hidden Cause of Arthritis in Danish Patients?
Status: Not yet recruiting | Type: Observational
Sponsor: Fredrikke Christie Knudtzen (Other)
Collaborators: Odense University Hospital (Other); Slagelse Hospital (Other); Gødstrup Hospital (Other); Aalborg University Hospital (Other); Regionshospitalet Silkeborg (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Vejle Hospital (Other); Frederiksberg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Fredrikke Christie Knudtzen, MD, Specialist in Infectious Diseases, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: S-20240040
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lyme Arthritis
Keywords: Lyme arthritis; Borrelia arthritis; Borreliosis; Monoarthritis; Oligoarthritis
MeSH Terms: conditions — Lyme Disease; Borrelia Infections; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — For each patient, blood samples and synovial fluid from joints with arthritis will be retained in a biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with mono/oligoarthritis: All patients 18 years or older presenting at 8 rheumatological departments across Denmark with oligo/monoarthritis between 1.1.26-31.12.27.
  Interventions: Diagnostic Test: Synovial fluid Borrelia burgdorferi PCR

INTERVENTIONS:
Diagnostic Test: Synovial fluid Borrelia burgdorferi PCR — All patients will have a pan-Borrelia burgdorferi PCR performed on synovial fluid from joints with arthritis. The PCR-positive patients will be deemed to have Borrelia arthritis, all other patients will be deemed as not having Borrelia arthritis.

SUMMARY:
Why is this study being done? Borrelia arthritis is a joint infection caused by Borrelia bacteria transmitted by tick bites. It often affects the knee and can cause prolonged pain and swelling if not diagnosed and treated in time. While well recognized in North America, Borrelia arthritis is considered rare in Europe. Recent findings from the investigators in Denmark suggest it may be more common than previously thought and frequently diagnosed late.

The aim of this study is to improve knowledge about how often Borrelia arthritis occurs in Denmark, how it presents, how long diagnosis takes, and how patients recover. This may help ensure faster diagnosis and better treatment for future patients.

Who can take part? Patients referred to an including rheumatology department with inflammation in one or a few joints (mono- or oligoarthritis) may be invited to participate.

What does participation involve?

If a patient choose to participate:

* A blood sample will be taken to test for antibodies against Borrelia.
* Fluid from the affected joint(s) will be tested for Borrelia DNA.
* Blood and joint fluid samples will be stored in a secure research biobank for future analyses related to this study.
* The patient will complete a questionnaire about symptoms, health history, possible tick exposure, and the diagnostic process.
* Relevant information from the patients medical record (tests, treatments, and outcomes) will be collected.

All procedures are part of standard clinical care or involve minimal additional testing.

How will the information be used?

The study will investigate:

* How common Borrelia arthritis is among patients with joint inflammation in Denmark.
* Differences in symptoms, test results, diagnostic delays, treatment, and outcomes between patients with Borrelia arthritis and other forms of arthritis.

Risks and benefits Risks are minimal and mainly related to routine blood sampling and joint aspiration. The patient may not benefit directly, but the results may improve care for future patients.

Confidentiality and voluntary participation All personal data will be handled confidentially according to data protection regulations. Participation is voluntary, and patients may withdraw at any time without affecting their medical care.

Study period The study runs from January 1, 2026, to December 31, 2027 and includes patients from eight hospitals in Denmark.

DETAILED DESCRIPTION:
Introduction Borrelia arthritis is, despite being a painful and debilitating disease, barely studied in Europe. The investigating research group has discovered an alarming number of cases in the last few years, and believe Borrelia arthritis is underdiagnosed in Denmark. This project therefore aims to systematically investigate the prevalence and trajectory of Borrelia arthritis in Denmark, in order to enhance the diagnostic capabilities, to improve outcomes for future patients, as well as reduce the costs for the Danish health care system.

Background Clinical aspect & outcome of Borrelia arthritis. Borrelia arthritis is a joint infection caused by the Borrelia burgdorferi bacteria group. Patients with Borrelia arthritis typically present months after tick exposure, most commonly with monoarthritis of the knee, although oligoarthritis can occur. Diagnosing Borrelia arthritis has been a challenge, based solely on patient history and the presence of Borrelia IgG antibodies in plasma. Tools like polymerase chain reaction (PCR) analysis of synovial fluid provide better diagnostic accuracy, but are not readily available. Though antibiotic therapy relieves symptoms in most cases, Borrelia bacteria within the joint can activate the immune system leading to persistent synovial inflammation. In these patients, disease-modifying anti-rheumatic drugs are required, and recovery may take months to years, with risk of lasting pain and disability.

Distribution & prevalence. In North America, Borrelia arthritis is found in 30% of Lyme borreliosis cases, whereas in Europe, it is considered rare. This discrepancy is attributed to differences in Borrelia species and their tissue tropism: European species tend to primarily affect the skin and nervous system, while American species more commonly target the joints. Current knowledge on European Borrelia arthritis epidemiology and outcomes is limited, but it is thought to present with subtler symptoms than in North America, potentially leading to overlooked cases. A French cohort study reported a median delay of 5 months from symptom onset to diagnosis, and found several Borrelia-species involved. Few studies have been conducted in Scandinavia. In Southern Norway a study found the Borrelia arthritis incidence to be 2.7/100,000 adults, while it was 2.3% in a high-endemic area of Sweden. In Denmark, a registry study in the Capital Region found that 4 of 146 patients with Borrelia antibodies had a possible Borrelia arthritis.

Current status in Denmark. Since 2021, the investigators research group has identified multiple patients with Borrelia arthritis from a specific area (Marbæk plantage) near Esbjerg. This indicates an emerging Borrelia-hotspot in this area, possibly an effect of climatic changes on the distribution of Borrelia host animals and tick abundance. Initially, Borrelia arthritis was not suspected in these cases, but as awareness of the disease increased, the diagnostic delay was reduced: from 38 months in the first patient to six weeks in the most recent one. With heightened attention on the condition and with the availability of improved diagnostic tools, more than 50 additional cases of Borrelia arthritis from other regions of Denmark have been identified since 2023. The high positive sample rate of 49% (25 of 51 patients tested so far in 2025) suggests undertesting and overlooked cases.

Aim. More knowledge regarding the incidence and clinical features of Borrelia arthritis in Denmark is needed, to ensure a timely and appropriate diagnosis and treatment, thereby reducing risk of complications for affected patients in the future. With this project, the aim is to determine the incidence of Borrelia arthritis in patients with mono/oligoarthritis across all Danish regions, to characterize the clinical presentation of Borrelia Arthritis in Northern European patients, and to determine if the Borrelia-species involved belong to genotypes associated with Borrelia arthritis in North America or the more common European types.

Hypotheses. The investigators hypothesise that Borrelia arthritis is an underrecognised infection in Denmark, and that Borrelia arthritis has a favourable prognosis compared with other causes of mono/oligoarthritis, that Borrelia arthritis is an emerging infection in Northern Europe due to climate changes favoring tick survival, and that the Borrelia genotypes responsible for Northern European Borrelia arthritis differ from Northern American strains.

Methods Sub-study 1 - Borrelia arthritis incidence & outcome study: To establish the number of Borrelia arthritis cases, all patients presenting with mono/oligoarthritis at the Departments of Rheumatology at eight hospitals across Denmark will be tested prospectively with a serum-Borrelia IgG antibody test from 1.1.26 until 31.12.27. All patients will have their synovial fluid tested for B.burgdorferi DNA by PCR and sampled blood and synovial fluid tested for intrasynovial synthesis of B.burgdorferi antibodies. A biobank will be established at the Department of Clinical Microbiology, OUH, containing blood and synovial fluid. Around 25 patients from each of the eight sites are expected to be included yearly, in all 350-400 patients in two years. A RedCap database will be established including data on 1-year arthritis outcomes where the patients with Borrelia arthritis and patients with arthritis of other origin will be compared.

Sub-study 2 - Borrelia arthritis characterisation study: A questionnaire for all patients included in Study 1 will be designed. The RedCap database will include data from the questionnaire and from patient charts; demographic information, clinical history (symptom debut, affected joints), course of disease (fluctuating, stable or progressing arthritis, pain, fever, other symptoms, and comorbidities), tick exposure history, diagnostic pathway (health professionals involved), diagnostic test results (joint fluid (WBC count, direct microscopy, culture, PCR), blood tests (Borrelia antibody status, hematology, inflammatory markers, uric acid, autoantibodies), final diagnosis and treatment (pain medicine, anti-inflammatory drugs and antibiotics). The investigators will compare the Borrelia arthritis patients (cases) with the arthritis patients without Borrelia (control group) in terms of tick-bite history and exposure, symptoms and paraclinical data through statistical analyses.

Expected impact. The primary expected outcome is an improved understanding of the occurence, clinical characteristics, and microbiological profile of Borrelia arthritis. By collecting comprehensive data on diagnostic pathways and outcomes, the research will provide insights into the challenges faced by Borrelia arthritis patients, especially in the context of delayed diagnoses. The study's findings will inform targeted interventions, including the development of more efficient diagnostic protocols and increased awareness among healthcare providers regarding symptoms and diagnostic markers of Borrelia arthritis. Additionally, the establishment of a biobank will facilitate future research into the disease's pathophysiology and guide the development of tailored treatment strategies. Ultimately, the study could lead to the establishment of public health initiatives aimed at better prevention, early detection, and management of Borrelia arthritis in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Presenting with mono/oligoarthritis at one of the including Departments of Rheumatology between 1/1-26 and 31/12-27
* Danish abilities to read and consent to inclusion
* Oral and written consent including biobank

Exclusion Criteria:

* Diagnoses of other inflammatory arthritis in relation to current arthritis episode (gout, pseudo-gout, rheumatoid arthritis, psoriatic arthritis, peripheral spondyloarthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to one of 8 Rheumatological departments: Aalborg, Gødstrup, Silkeborg, Esbjerg, Vejle, Odense, Slagelse or Frederiksberg Hospital within the studyperiod.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Sub-study 1: 1-year cure rate Borrelia arthritis vs. control group | 1 year after inclusion
  Number of patients recovered drug-free (antibiotic treatment and/or DMARDs) one year after inclusion, in the Borrelia arthritis group and in the control group. Difference between the groups.
Sub-study 2: Serum-Borrelia IgG antibodies | At study inclusion
  Statistical difference between the 2 groups (Borrelia arthritis vs. control group) at baseline of number of patients with a serum-Borrelia IgG antibody.

SECONDARY OUTCOMES:
Sub-study 1: Borrelia arthritis incidence and Borrelia burgdorferi genospecies | At study inclusion
  Proportion of all included patients with a Bb PCR positive joint fluid, and classification of the B. burgdorferi strains found in synovial fluid of patients with Borrelia arthritis.
Sub-study 1: 6-month cure rate Borrelia arthritis vs. control group | 6 months after study inclusion
  Number of patients recovered drug-free (antibiotic treatment and/or DMARDs) six months after inclusion, in the Borrelia arthritis group and in the control group. Difference between the groups.
Sub-study 2: Difference between groups in which joints are affected | At study inclusion
  Statistical difference between the two groups at baseline in joints involved (knee, ankle, hip, shoulder, elbow, other) and number of joints involved (1, 2, 3 or more)
Sub-study 2: Difference between groups in amount of synovial fluid. | At study inclusion
  Statistical difference between the two groups at baseline in estimated ml of synovial fluid in ml in affected joints

OTHER OUTCOMES:
Age | At study inclusion
  Difference ibetween the 2 groups in median age at date of inclusion
Sex | At study inclusion
  Difference between the 2 groups in % male sex.
Number of tick-bites 1 year | At study inclusion
  Difference in the 2 groups between number of tick-bites in the last year up to date of inclusion
Number of tick-bites last 5 years | At study inclusion
  Difference in the 2 groups between number of tick-bites in the last year and in the last 5 years leading up to inclusion.
Tick-bite risk behaviour | At study inclusion
  Difference in the 2 groups in number of patients with risk behaviour (hiking, hunting, scouts, orienteers, golfing, extensive gardening)
Arthritis presentation | At study inclusion
  Difference between the 2 groups in arthritis presentation (continuous or relapsing/remitting).
DAS 28 score | At study inclusion and again at 6 month follow-up control and 1 year follow-up control
  Difference between the 2 groups in calculated DAS 28 score. Calculated from the following variables: Tender Joint Count 28 score, Swollen Joint Count 28 score, C-reactive protein (mg/L) and Global VAS score (score from 0-100) with this calculation: (0.56*sqrt([tj_count])) + (0.28*sqrt([sj_count])) + (0.014*[global_vas]) + (0.36*log([crp] + 1)) + 0.96
BMI | At study inclusion
  Difference between the 2 groups in Body Mass Index, calculated by (Weight in kg / (Height in cm)²) x 10,000
Comorbidities | At study inclusion
  Differences in comorbidities in the last 5 years before study inclusion, using the Charlson comorbidity index, with following groups; score of 0, score of 1, score of 2, and score of >2.
BRAF score | At study inclusion and again at 6 months and 1 year follow up.
  Differences between the groups in BRAF score, testing for fatigue.
Anti-CCP | at study inclusion
  Difference between groups in number of patients with a positive (5-15 kU/L) or highly positive (>15 kU/L) S- anti-cyclic citrullinated protein (kU/L)
Rheumatoid factor | At study inclusion
  Difference between the 2 groups in number of patients with a positive S-Rheumatoid factor

CONTACTS AND LOCATIONS:
Overall Officials: Fredrikke C Knudtzen, MD, Principal Investigator — Odense University Hospital, Department of Infectious Diseases

IPD SHARING:
Plan to Share IPD: No
Due to Danish GDPR rules we do not plan on making IPD data available to other researchers. However, the sponsor-investigator responsible for the study can be contacted by interested parties.

REFERENCES:
- [Background] Unlu AM, Andersen NS, Larsen SL, Skarphedinsson S, Chrysidis S, Knudtzen FC, Lage-Hansen PR. Differentiating Lyme arthritis: a case-based review. Rheumatol Int. 2024 Nov;44(11):2671-2678. doi: 10.1007/s00296-024-05618-0. Epub 2024 May 25. PMID 38795123
- [Background] Arvikar SL, Steere AC. Diagnosis and treatment of Lyme arthritis. Infect Dis Clin North Am. 2015 Jun;29(2):269-80. doi: 10.1016/j.idc.2015.02.004. PMID 25999223
- [Background] Tory HO, Zurakowski D, Sundel RP. Outcomes of children treated for Lyme arthritis: results of a large pediatric cohort. J Rheumatol. 2010 May;37(5):1049-55. doi: 10.3899/jrheum.090711. Epub 2010 Apr 1. PMID 20360182
- [Background] Corre C, Coiffier G, Le Goff B, Ferreyra M, Guennic X, Patrat-Delon S, Degeilh B, Albert JD, Tattevin P. Lyme arthritis in Western Europe: a multicentre retrospective study. Eur J Clin Microbiol Infect Dis. 2022 Jan;41(1):21-27. doi: 10.1007/s10096-021-04334-y. Epub 2021 Aug 20. PMID 34417687
- [Background] Steere AC. Treatment of Lyme Arthritis. J Rheumatol. 2019 Aug;46(8):871-873. doi: 10.3899/jrheum.190320. No abstract available. PMID 31371661
- [Background] Steere AC, Angelis SM. Therapy for Lyme arthritis: strategies for the treatment of antibiotic-refractory arthritis. Arthritis Rheum. 2006 Oct;54(10):3079-86. doi: 10.1002/art.22131. No abstract available. PMID 17009226
- [Background] Stanek G, Reiter M. The expanding Lyme Borrelia complex--clinical significance of genomic species? Clin Microbiol Infect. 2011 Apr;17(4):487-93. doi: 10.1111/j.1469-0691.2011.03492.x. PMID 21414082
- [Background] Cerar T, Strle F, Stupica D, Ruzic-Sabljic E, McHugh G, Steere AC, Strle K. Differences in Genotype, Clinical Features, and Inflammatory Potential of Borrelia burgdorferi sensu stricto Strains from Europe and the United States. Emerg Infect Dis. 2016 May;22(5):818-27. doi: 10.3201/eid2205.151806. PMID 27088349
- [Background] Haugeberg G, Hansen IJ, Skarpaas T, Noraas S, Kjelland V. Lyme arthritis in Southern Norway--an endemic area for Lyme borreliosis. BMC Infect Dis. 2014 Apr 5;14:185. doi: 10.1186/1471-2334-14-185. PMID 24708707
- [Background] Berglund J, Hansen BU, Eitrem R. Lyme arthritis--a common manifestation in a highly endemic area in Sweden. J Rheumatol. 1995 Apr;22(4):695-701. PMID 7791166
- [Background] Muller T, Locht H, Panum I, Nielsen L, Jensen B. Lyme arthritis is rare in Eastern Denmark. Dan Med J. 2021 Oct 26;68(11):A05210423. PMID 34983732